CLINICAL TRIAL: NCT06089265
Title: Short-term Safety and Efficacy of Ketohexokinase Inhibition in Patients With Hereditary Fructose Intolerance
Brief Title: Ketohexokinase Inhibition in Hereditary Fructose Intolerance
Acronym: KHKi in HFI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83631.068.23 / METC23-006
Record Dates: First submitted 2023-05-15; First posted 2023-10-18 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: HFI

STUDY DESIGN:
Intervention Model Description: open label, pilot study
Masking Description: all HFI participants will get the medication, no placebo will be used. Controls will get no medication or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFI patients (Experimental): HFI participants will receive PF-06835919 for 9 days. Dosage; once daily 300 mg PF-06835919 in the form of 3 tablets, oral.
  Interventions: Drug: PF-06801591
- Healthy controls (No Intervention): Healthy controls will receive no intervention, but a single fructose tolerance test.

INTERVENTIONS:
Drug: PF-06801591 — Active ketohexokinase inhibitor
  Other Names: KHKi
  Arms: HFI patients

SUMMARY:
Hereditary fructose intolerance (HFI) is a rare inborn error of metabolism. Patients with HFI develop acute abdominal pain, nausea, vomiting, hypoglycemia and proximal tubular dysfunction upon consumption of a fructose containing food product. In rare cases, (prolonged) fructose consumption can even lead to liver and kidney failure. Patients with HFI are therefore treated with a lifelong fructose-restricted diet. Animal studies have shown that the clinical manifestations of HFI are abrogated upon inhibition of ketohexokinase (KHK), the enzyme that catalyses the first step in fructose metabolism.

Recently, PF-06835919, a KHK inhibitor (KHKi), was developed as a new treatment for non-alcoholic fatty liver disease. The compound was well tolerated in several phase II clinical trials.

It is hypothesized that PF-06835919 is also effective in patients with HFI.

DETAILED DESCRIPTION:
Rationale: Hereditary fructose intolerance (HFI) is a rare inborn error of metabolism. Patients with HFI develop acute abdominal pain, nausea, vomiting, hypoglycemia and proximal tubular dysfunction upon consumption of a fructose containing food product. In rare cases, (prolonged) fructose consumption can even lead to liver and kidney failure. Patients with HFI are therefore treated with a lifelong fructose-restricted diet. Animal studies have shown that the clinical manifestations of HFI are abrogated upon inhibition of ketohexokinase (KHK), the enzyme that catalyses the first step in fructose metabolism.

Recently, PF-06835919, a KHK inhibitor (KHKi), was developed as a new treatment for non-alcoholic fatty liver disease. The compound was well tolerated in several phase II clinical trials.

It is hypothesized that PF-06835919 is also effective in patients with HFI. Objective: To study the effects of PF-06835919 on fructose tolerance and intrahepatic lipid content in patients with HFI. Study design: open-label, pilot study Study population: three adult patients with HFI will be treated with PF-06835919. Five adult healthy individuals will be included (but not be treated) as a reference. Intervention (if applicable): Patients receive once daily (in the morning) three tablets of 100 mg PF-06835919 for 9 days. They will subsequently be gradually exposed to increasing doses of either oral fructose or glucose (in a blinded fashion). Healthy individuals will only undergo oral fructose exposure, as a reference. Main study parameters/endpoints: Intrahepatic lipid content assessed by proton magnetic resonance spectroscopy (at baseline and completion), intestinal fructose tolerance (after oral fructose in comparison to oral glucose), hepatic fructose tolerance (serum glucose and phosphate after oral fructose in comparison to healthy individuals) and renal fructose tolerance (urinary glucose, phosphate, pH and amino acids after oral fructose in comparison to healthy individuals). Nature and extent

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to provide signed and dated written informed consent prior to any study specific procedures
* Use of effective contraception (only applicable to premenopausal women; a pregnancy test will be performed in these women at baseline)
* Aged ≥ 18 years

Exclusion Criteria:

* Diabetes mellitus
* Pregnancy
* Patients with congestive heart failure and/or severe renal and or liver insufficiency
* Uncontrolled hypertension
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the investigator which would possibly hamper our study results
* Use of drugs that inhibit organic anion transporting polypeptide B1 (OATPB1) transporters (e.g. rifampicin, gemfibrozil, ciclosporine, erythromcyin and clarithromycin)*
* Treatment with irinotecan* Any contra-indications for MRI scanning*
* Subjects who do not want to be informed about unexpected medical findings

  * Exclusion criterion for HFI patients only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Intestinal Fructose tolerance, | 9 days
  a visual analog scale from 1-10 for abdominal pain will be used. Additional every 5 minutes the participant will be asked if he/she is nauseous, and more, less or similar nauseous as 5 minutes before.
Intestinal Fructose tolerance, | 9 days
  Every 5 minutes the participant will be asked if he/she is nauseous, and more, less or similar nauseous as 5 minutes before.
Renal Fructose tolerance | 9 days
  Urinary pH
Renal Fructose tolerance | 9 days
  Glucose content, mmol/L
Renal Fructose tolerance | 9 days
  Phosphate content mmol/L
Renal Fructose tolerance | 9 days
  Amino acid content mmol/L
Hepatic fructose tolerance | 9 days
  Serum glucose levels, mmol/L
Hepatic fructose tolerance | 9 days
  Serum phosphate levels, mmol/L

SECONDARY OUTCOMES:
Intrahepatic lipid content | 9 days
  measured using 1H-MRS at baseline and completion
Blood pressure | 9 days
  measured at baseline and completion. Both systolic and diastolic pressure will be assessed
Glycosylated transferrin | 9 days
  measured at baseline and completion.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data can be obtained with the PI on request